CLINICAL TRIAL: NCT05648318
Title: 1L Oral Lactulose is an Effective Regimen for Bowel Preparation in Low-risk Patients
Brief Title: Comparison of Oral Lactulose Versus Polyethylene Glycol for Bowel Preparation in Low-risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhang Xiaofeng,MD (Other)
Responsible Party: Sponsor-Investigator, Zhang Xiaofeng,MD, chief physician, First People's Hospital of Hangzhou
Organization: First People's Hospital of Hangzhou (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 20211206301
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Colonic Neoplasms
Keywords: colonoscopy; bowel preparation
MeSH Terms: conditions — Colonic Neoplasms | interventions — Lactulose

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactulose oral solution (LOS) (Experimental)
  Interventions: Drug: Lactulose oral solution
- polyethylene glycol (PEG) (Active Comparator)
  Interventions: Drug: PEG

INTERVENTIONS:
Drug: Lactulose oral solution — In the LOS group, patients were instructed to drink 200ml lactulose (Duphalac, Olst, the Netherlands; 200ml/bottle) diluted with clear water into 1L 4-6h before colonoscopy at a rate of 250ml every 30min.
  Arms: Lactulose oral solution (LOS)
Drug: PEG — patient in the PEG group were instructed to drink 2L of PEG (each liter containing 59g PEG 4000, 1.46g sodium chloride, 5.68g sodium sulfate, 0.74g potassium chloride, 1.68g sodium bicarbonate; WanHe Pharmaceutical Co, Ltd., China) 4-6h before colonoscopy at a rate of 250ml every 15min
  Arms: polyethylene glycol (PEG)

SUMMARY:
Adequate quality of bowel preparation(BP) is essential for colonoscopy. In recently, Kang suggested that for low-risk patients, single dose of 2L PEG is an effective regimen for bowel preparation.However, due to the poor palatability, there still more than 30% patients with 2L regimen experienced nausea or vomiting in our center.

Oral lactulose is a treatment for constipation. Several studies have compared the effectiveness between use PEG and lactulose for colonoscopy preparation in average-risk patients. However, the data in low-risk patients is vacant. The objective of current study was to compared the effectiveness of bowel preparation and patient tolerance using lactulose and 2L PEG regimen in low-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old and with low-risk were eligible. Patients were considered as low risk if they did not meet any of the following risk factors: age>70 years old, body mass index (BMI)>25Kg/m2, constipation, Parkinson's disease, diabetes, history of stroke or spinal cord injury, use of tricyclic antidepressant or narcotics.

Exclusion Criteria:

* (1) history of colorectal resection; (2) Known or suspected colonic stricture or obstructing tumor; (3) Known or suspected colonic perforation; (4) toxic colitis or megacolon; (5) use of prokinetic agents or purgatives within 7 days; (6) hemodynamic instability; (7) pregnancy or lactation; (8) inability to provide informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Bowel preparation | 1hour
  Boston bowel preparation score (BBPS)：cleanliness of each part of the colon: 0=unprepared colon segment with mucosa not seen because of solid stool that cannot be cleared; 1=portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen because of staining, residual stool, and/or opaque liquid; 2=minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well; 3=entire mucosa of colon segment seen well with no residual staining, small fragments of stool, or opaque liquid.

SECONDARY OUTCOMES:
Adverse events | 1hour
Willingness to repeat bowel preparation | 1hour
  We will ask patients in the form of questionnaire whether they are willing to repeat the same bowel preparation method if they need colonoscopy examination again
Adenoma detection rate | 7 days
Cecal intubation rate | 1hour
insertion time | 1hour
withdrawal time | 1hour

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zhang, MD, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou first people's Hospital, Hangzhou, Zhejiang, China